CLINICAL TRIAL: NCT04611191
Title: The Effect of Team Sports on the Susceptibility to Thrombosis in Elderly Men and Women in a Municipality Setting
Brief Title: The Effect of Team Sports on the Risk of Thrombosis in Elderly Individuals in a Municipality Setting (TEAM-AGE)
Acronym: TEAM-AGE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Swansea University (Other)
Responsible Party: Principal Investigator, Ylva Hellsten, Professor, University of Copenhagen
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Team sports and thrombosis
Record Dates: First submitted 2020-10-26; First posted 2020-11-02 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Thrombosis; Exercise Training; Sex Differences
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Team Sports (Experimental): Elderly men and women performing team sports in local sports clubs
  Interventions: Other: Team Sports
- Control (Experimental): Elderly men and women continue their normal lifestyle
  Interventions: Other: Control

INTERVENTIONS:
Other: Team Sports — The intervention involves team sports in sports clubs in local municipalities
  Arms: Team Sports
Other: Control — The intervention involves a control condition with participants continuing their normal way of living
  Arms: Control

SUMMARY:
Cardiovascular disease, and especially myocardial infarction, is the most common cause of death globally, and is particularly common in older individuals. Practical measures that can reduce both the prevalence and incidence of cardiovascular disease are of great value. It is well known that regular physical activity has a protective effect against the development of cardiovascular diseases such as acute myocardial infarction. It has been shown that physical activity can improve the function of the heart and blood vessels, but it is less well known how physical activity can affect the risk of formation of dangerous blood clots, and thus the risk of heart attack and stroke.

In a cross-sectional study it has been shown that a physically active lifestyle can reduce the risk of blood clot formation, but experimental evidence for the importance of a period of physical activity for the risk of blood clot formation is lacking. New methods have been set up for measuring the coagulation profile. The analyzes are performed on a blood sample and allow a thorough determination of platelet reactivity as well as an innovative measure of how the microstructure of a possible blood clot would develop. In this project, these methods is used to examine how physical activity, in the form of team sports, affects the coagulation profile of elderly men and women.

The increasing age-related risk of cardiovascular disease is associated with endothelial dysfunction and decrease in capillary density, and it has been shown that initiation of capillary growth is a successful method to treat cardiovascular disease. Therefore, this project will also investigate how a longer period of physical activity, in the form of team sports, affects capillary density and endothelial function in men and women aged 60-70 years. Both men and women will be recruited, as it is still unknown whether men and women respond differently to physical activity in relation to coagulation profile, susceptibility to blood clots and capillary density.

DETAILED DESCRIPTION:
Cardiovascular disease, and especially myocardial infarction, is the most common cause of death globally, and is particularly common in older individuals. Practical measures that can reduce both the prevalence and incidence of cardiovascular disease are of great value. It is well known that regular physical activity has a protective effect against the development of cardiovascular diseases such as acute myocardial infarction. Therefore, the American Heart Association also recommends ≥ 30 min. per day five days a week. It has been shown that physical activity can improve the function of the heart and blood vessels, but it is less well known how physical activity can affect the risk of formation of dangerous blood clots, and thus the risk of heart attack and stroke.

In a cross-sectional study it has been shown that a physically active lifestyle can reduce the risk of blood clot formation, but experimental evidence for the importance of a period of physical activity for the risk of blood clot formation is lacking. New methods have been set up for measuring the coagulation profile. The analyzes are performed on a blood sample and allow a thorough determination of platelet reactivity as well as an innovative measure of how the microstructure of a possible blood clot would develop. In this project, these methods is used to examine how physical activity, in the form of team sports, affects the coagulation profile of elderly men and women.

The increasing age-related risk of cardiovascular disease is associated with endothelial dysfunction and decrease in capillary density, and it has been shown that initiation of capillary growth is a successful method to treat cardiovascular disease. Therefore, this project will also investigate how a longer period of physical activity, in the form of team sports, affects capillary density and endothelial function in men and women aged 60-70 years. Both men and women will be recruited, as it is still unknown whether men and women respond differently to physical activity in relation to coagulation profile, susceptibility to blood clots and capillary density.

Part of the novelty of this present study consist of 1) linking the clinical measurements with data on sickness absence, disease development, etc. and with data on the underlying mechanisms, 2) examining the short-term effect (16 weeks) and the long-term effect (up to 2 years) of physical activity, in the form of team sports in a municipality setting, on coagulation, risk of blood clots, capillarization and endothelial function in general in the elderly, as well as 3) investigate whether there is a difference in the aforementioned measurements in men and women.

ELIGIBILITY:
Inclusion Criteria:

* Age: 60-70 years
* Physical activity ≤ 2 hours per week (except transportation by bike or by walking)
* BMI ≤ 30

Exclusion Criteria:

* Age <60 years
* Injuries that prevent the performance of team sports
* Participation in other clinical projects
* Smokes or has smoked within the last 10 years
* On hormone therapy (women)
* Not entered menopause (women)
* Has chronic diseases that are not expected, cf. the groups sought. Including heart problems, atrial fibrillation, cancer, immune diseases and previous strokes with functionally significant sequelae
* Being treated with oral steroids
* Has alcohol / drug abuse or is being treated with disulfiram (Antabus)
* Is unable to understand the contents of the document with informed consent or the experimental procedures

Ages: 60 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-12-30 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in clot microstructure in elderly individuals after 16 weeks and 1 year of team sports in local sports clubs, respectively | 12 months
  Clot microstructure is measured in a rheometer using unaltered whole blood
Changes in platelet reactivity in elderly individuals after 16 weeks and 1 year of team sports in local sports clubs, respectively | 12 months
  Platelet reactivity is measured with Light Transmission Aggregometry using platelet rich and platelet poor plasma
Plasma concentration of coagulation factors in elderly individuals after 16 weeks and 1 year of team sports in local sports clubs, respectively | 12 months
  Coagulation factors II, VII, X, VIII, D-dimer, fibrinogen and thrombin
Changes in capillary density in elderly individuals after 16 weeks and 1 year of team sports in local sports clubs, respectively | 12 months
  Capillary density will be assessed by histochemistry
Changes in proliferative capacity of endothelial cells from skeletal muscle biopsies in elderly individuals after 16 weeks and 1 year of team sports in local sports clubs, respectively | 12 months
  From a biopsy sample we isolate endothelial cells and run a proliferation assay

SECONDARY OUTCOMES:
Changes in blood pressure after 16 weeks and 1 year of team sports in local sports clubs, respectively, in elderly individuals | 12 months
  In a subgroup, blood pressure (systolic blood pressure, diastolic blood pressure and mean arterial pressure) will be measured at home with an automated blood pressure device.
Changes in maximal oxygen uptake after 16 weeks and 1 year of team sports in local sports clubs, respectively, in elderly individuals | 12 months
  Maximal oxygen uptake will be measured using a metabolic cart. The test protocol will be performed on a cycle ergometer using an incremental step test.
Changes in bodt composition after 16 weeks and 1 year of team sports in local sports clubs, respectively, in elderly individuals | 12 months
  Dual-energy x-ray absorptiometry (DXA) is used to determine fat free mass, fat mass as well as bone mineral content. These values will be presented in absolute (g) as well as relative values (percentage)

CONTACTS AND LOCATIONS:
Overall Officials: Jens Bangsbo, Dr.Sci., Principal Investigator — Nutrition, Exercise and Sports, 2200 Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No